CLINICAL TRIAL: NCT04581954
Title: Randomised Multi-arm Trial of Ruxolitinib (RUX) and Fostamatinib (FOS) for COVID-19 Pneumonia
Brief Title: Inflammatory Signal Inhibitors for COVID-19 (MATIS)
Acronym: MATIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Rigel Pharmaceuticals (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20HH5926; 2020-001750-22 (EudraCT Number)
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Coronavirus; Covid19; Pneumonia
Keywords: coronavirus; covid19; pneumonia; ruxolitinib; fostamatinib
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Pneumonia | interventions — ruxolitinib; fostamatinib; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of care (Active Comparator)
  Interventions: Other: Standard of care
- Fostamatinib (Active Comparator)
  Interventions: Drug: Fostamatinib
- Ruxolitinib (Active Comparator)
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is a Janus kinase 1 (JAK1)/Janus kinase 2 (JAK2) inhibitor approved for clinical use in the treatment of splenomegaly, myelofibrosis, polycythaemia vera and graft-versus-host disease. It is an oral agent with a rapid mode of action.
  Arms: Ruxolitinib
Drug: Fostamatinib — Fostamatinib is a tyrosine kinase inhibitor with activity against spleen tyrosine kinase (SYK). It has approved for the treatment of thrombocytopenia in adult patients with chronic immune thrombocytopenia (ITP).
  Arms: Fostamatinib
Other: Standard of care — Standard of care treatment as per site-level policies and guidelines.
  Arms: Standard of care

SUMMARY:
The Multi-arm trial of Inflammatory Signal Inhibitors for COVID-19 (MATIS) study is a two-stage, open-label, randomised controlled trial assessing the efficacy of ruxolitinib (RUX) and fostamatinib (FOS) individually, compared to standard of care in the treatment of COVID-19 pneumonia. The primary outcome is the proportion of hospitalised patients progressing from mild or moderate to severe COVID-19 pneumonia. Patients are treated for 14 days and will receive follow-up assessment at 7, 14 and 28 days after the first study dose. Patients with mild or moderate COVID-19 pneumonia will be recruited. Initially, n=171 (57 per arm) patients will be recruited in Stage 1. Following interim analysis to assess the efficacy and safety of the treatments, approximately n=285 (95 per arm) will be recruited during Stage 2.

DETAILED DESCRIPTION:
COVID-19 pneumonia is characterised by respiratory and multi-organ failure in the context of marked systemic inflammation. It is caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARSCoV2) infection. The hallmark of severe disease is hypoxia and a radiological pattern of acute lung injury that shares features with Acute Respiratory Distress Syndrome (ARDS). Early features of COVID-19 result from host viral response and typically include symptoms such as fever and dry cough. Later features, typically occurring beyond 7 days, are characterised by marked and progressive systemic inflammation, identified by elevations in a plethora of inflammatory molecules such as C-reactive protein, ferritin and IL6. In a subset of patients, hyperinflammatory responses drive acute lung injury and may result in catastrophic multi-organ failure and death.

The aetiology of COVID-19 induced ARDS is incompletely understood but appears to be associated with lung inflammation effected by a monocytic and neutrophilic infiltration, elevated cytokine levels and tissue damage. Elevations in circulating inflammatory molecules are associated with poor prognosis. In particular, the COVID-19 hyperinflammatory response syndrome is associated thrombotic complications which are postulated to drive cardiac dysfunction and microvascular thrombi, suggested by elevations in troponin and D-dimer, respectively. Similar hyperinflammatory responses are also seen in macrophage activation syndromes such as haemophagocytic lymphohistiocytosis, or in the cytokine release syndrome associated with chimeric antigen receptor T cell therapy. Further, preliminary data from China and Italy have shown immediate resolution of symptoms using anti-interleukin-6 agents (anti-IL6) therapy and Janus kinase inhibitors (JAK)/signal transducer and activator of transcription (STAT) inhibitors in patients with severe disease. There may be an early window of opportunity to treat the COVID-19 hyperinflammatory syndrome before acute lung injury leads to organ failure.

There are currently no approved treatments for COVID-19 pneumonia. This is a protocol for a randomised controlled, multi-arm trial of early intervention with inflammatory signal inhibitors.

Study purpose

A number of therapeutic interventions targeting inflammatory signalling might reduce the severity of the inflammatory response phase resulting in amelioration of the lung damage thereby averting respiratory failure and the need for mechanical ventilation. This trial aims to evaluate the efficacy of two inhibitors of key signalling pathways using drugs which are already licensed for use in other clinical indications.

Primary objective

The primary objective is to determine the efficacy of RUX and FOS to reduce the proportion of hospitalised patients progressing from mild/moderate to severe COVID-19 pneumonia. A modified World Health Organization (WHO) COVID-19 Severity Ordinal Scale (COVID-19 Therapeutic Trial Synopsis published 18th February 2020) will be used to grade clinical deterioration from Hospitalised Mild Disease (<5) to Hospitalised Severe Disease (greater than or equal to 5). The modification includes an additional grade for Hospitalised Severe Disease that allows the capture of clinical deterioration in patients for whom escalation in organ support is not offered. Patients are eligible for recruitment to MATIS at grades 3 or 4. These patients stand to gain the greatest benefit from inflammatory signal inhibitors that may ameliorate the cytokine storm and prevent organ failure.

Secondary objectives

* Determine the efficacy of RUX or FOS to reduce mortality
* Determine the efficacy of RUX or FOS to reduce the need for invasive ventilation and/or ECMO
* Determine the efficacy of RUX or FOS to reduce the need for non-invasive ventilation including CPAP or high flow nasal oxygen
* Determine the efficacy of RUX or FOS to reduce the proportion of patients suffering clinically significant oxygen desaturation
* Determine the efficacy of RUX or FOS to reduce the need for renal replacement therapy
* Determine the efficacy of RUX and FOS to reduce the incidence of venous thromboembolism COVID-19 pneumonia
* Determine the efficacy of RUX and FOS to improve the severity of COVID19 pneumonia on a modified WHO COVID19 Ordinal Scale
* Determine the efficacy of RUX or FOS to reduce the level of inflammatory biomarkers
* Determine the efficacy of RUX or FOS to reduce blood ferritin, CRP, LDH and D-dimer
* Determine the efficacy of RUX or FOS to reduce the level of serum creatinine.
* Determine the efficacy of RUX or FOS to reduce duration of hospital admission

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥ 18 years at screening
* Patients with mild or moderate C19 pneumonia, defined as Grade 3 or 4 severity by the WHO COVID-19 Ordinal Scale by
* Patients meeting criteria: Hospitalization AND SARS-CoV2 infection (clinically suspected* or laboratory-confirmed) AND Radiological change consistent with COVID-19 disease
* C-reactive protein (CRP) greater than or equal to 30mg/L
* Informed consent from patient or personal or professional representative
* No medical history that might, in the opinion of the responsible clinician, put the patient at significant risk if he/she were to participate in the trial
* Agreement to abstain from sexual intercourse or use contraception that is >99% effective for all participants of childbearing potential for 42 days after the last dose of study drug. For male participants, agreement to abstain from sperm donation for 42 days after the last dose of study drug.
* Able to read English. Non-English speakers will be able to join the study. If patients are unable to understand verbal or written information in English - hospital translation services will be requested at the participating site for the participant where possible.

Exclusion Criteria:

* Requiring either invasive or non-invasive ventilation including CPAP or high flow nasal oxygen at any point after hospital admission and before baseline not related to a pre-existing condition (e.g. obstructive sleep apnoea)
* Grade ≥ 5 severity on the modified WHO COVID-19 Ordinal Scale, viz. O2 saturation < 90% on ≥ 60% inspired oxygen at baseline; non-invasive ventilation; or invasive mechanical ventilation at any point since hospital admission.
* In the opinion of the investigator, progression to death is inevitable within the next 24 hours, irrespective of the provision of therapy
* Known severe allergic reactions to the investigational agents
* Child Pugh B or C grade hepatic dysfunction
* Use of drugs within the preceding 14 days that are known to interact with any study treatment (FOS or RUX), as listed in the Summary of Product Characteristics
* Pregnant or breast feeding
* Any medical condition or concomitant medication that in the opinion of the investigator would compromise subjects' safety or compliance with study procedures.
* Any medical condition which in the opinion of the principal investigator would compromise the scientific integrity of the study
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Progression from mild to severe COVID-19 pneumonia within 14 days in hospitalised patients | Day 14
  Patients are recruited at a WHO COVID-19 Severity Score of 3 and 4 and the primary endpoint is the comparison of patients whose COVID-19 pneumonia progresses to a severity score ≥ 5 on the modified WHO Ordinal Scale. Specifically, the primary endpoint is met when the following are recorded within 14 days:
  * Death
  * Requirement for invasive ventilation
  * Requirement for non-invasive ventilation including CPAP or high flow nasal oxygen
  * O2 saturation < 90% on ≥60% inspired oxygen

SECONDARY OUTCOMES:
Mortality | Day 14
  all cause mortality
Mortality | Day 28
  all cause mortality
Invasive ventilation | Day 14
Invasive ventilation | Day 28
Non-invasive ventilation including CPAP and high flow nasal oxygen | Day 14
Non-invasive ventilation including CPAP and high flow nasal oxygen | Day 28
Renal replacement therapy | Day 14
Renal replacement therapy | Day 28
Venous Thromboembolism | Day 14
Venous Thromboembolism | Day 28
Serum Creatinine | Day 14
Serum Creatinine | Day 28
Length of stay | Day 28
Serious Adverse Events | Day 28
Serious Adverse Reactions | Day 28
Treatment discontinuation | Day 14
Change in severity from the modified WHO COVID-19 ordinal scale | Day 14
Change in severity from the modified WHO COVID-19 ordinal scale | Day 28
C-Reactive protein | Day 14
C-Reactive protein | Day 28
lactate dehydrogenase | Day 14
lactate dehydrogenase | Da 28
ferritin | Day 14
ferritin | Da 28
d-dimer | Day 14
d-dimer | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Nichola Cooper, Principal Investigator — Imperial College London
Locations (5):
- United Kingdom (5):
  - The Leeds Teaching Hospital - St James University Hospitals NHS Trust, Leeds
  - London North West University Healthcare, London
  - Imperial College Healthcare NHS Trust, London
  - Royal Berkshire NHS Foundation Trust, Reading
  - Sheffield Teaching Hospitals NHS Foundation Trust - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data (excluding free text fields) and supporting documentation (including the MATIS study protocol, Statistical Analysis Plan and data dictionary) can be made available upon reasonable request from the corresponding author (n.cooper@imperial.ac.uk) for the purposes of scientific research including secondary analysis of the data or for individual participant meta-analysis with appropriate human research ethics approvals and data transfer agreements in place

REFERENCES:
- [Derived] Hazell L, Pillay C, Cornelius V, Phillips R, Charania A, Wason J, Cherlin S, Savic S, Whittington A, Neelakantan P, Collini P, Cook L, Willicome M, Milojkovic D, Kon OM, Youngstein T, Innes A, Thursz M, Cooke GS, Vergis N, Cooper N. Multiarm multistage randomised controlled trial of inflammatory signal inhibitors (MATIS) for patients hospitalised with COVID-19 pneumonia during the UK pandemic. BMJ Open. 2026 Feb 5;16(2):e100583. doi: 10.1136/bmjopen-2025-100583. PMID 41644167
- [Derived] Vergis N, Phillips R, Cornelius V, Katsarou A, Youngstein T, Cook L, Willicombe M, Pilay C, Shturova T, Almonte M, Charania A, Turner R, Kon OM, Cooke G, Thursz M, Cherlin S, Wason J, Milojkovic D, Innes AJ, Cooper N. Multi-arm Trial of Inflammatory Signal Inhibitors (MATIS) for hospitalised patients with mild or moderate COVID-19 pneumonia: a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Apr 12;22(1):270. doi: 10.1186/s13063-021-05190-z. PMID 33845867

DOCUMENTS (2):
  • Study Protocol (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT04581954/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT04581954/SAP_001.pdf